CLINICAL TRIAL: NCT02981966
Title: Effect of Dapagliflozin on Hepatic and Renal Glucose Metabolism Subjects (11038)
Brief Title: Effect of Dapagliflozin on Hepatic and Renal Glucose Metabolism Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC20160596H
Record Dates: First submitted 2016-11-30; First posted 2016-12-05 (Estimated); Results first posted 2023-06-06 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- T2DM individuals on Dapagliflozin (Active Comparator): Individuals with type 2 diabetes mellitus - dapagliflozin
  Interventions: Drug: Dapagliflozin
- T2DM individuals on Placebo (Placebo Comparator): Individuals with type 2 diabetes mellitus on placebo
  Interventions: Drug: Placebo
- Normal Glucose Tolerance (NGT) on Dapagliflozin (Active Comparator): Individuals with normal glucose tolerance - dapagliflozin
  Interventions: Drug: Dapagliflozin
- Normal Glucose Tolerance (NGT) Placebo (Placebo Comparator): Individuals with normal glucose tolerance - on placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin — dapagliflozin, 10mg tablet
  Other Names: Farxiga
  Arms: Normal Glucose Tolerance (NGT) on Dapagliflozin; T2DM individuals on Dapagliflozin
Drug: Placebo — Placebo for dapagliflozin
  Arms: Normal Glucose Tolerance (NGT) Placebo; T2DM individuals on Placebo

SUMMARY:
Researchers hope to determine the organ (liver and/or kidney) responsible for the increase in endogenous glucose production (EGP) following the induction of glucosuria (when glucose is excreted in detectable amounts in the urine) with an SGLT2 inhibitor, dapagliflozin.

DETAILED DESCRIPTION:
Researchers will measure the rate of hepatic and renal glucose production following dapagliflozin administration to determine the site of increase in EGP, liver versus kidney. Researchers will measure the rate of whole body glucose production with 3-3H-glucose (a form of radioactive glucose) and renal glucose production by renal vein catheterization in T2DM (type 2 diabetes mellitus) and in lean healthy NGT (normal glucose tolerance) individuals. Because the increase in EGP is associated with an increase in plasma glucagon concentration and renal glucose production is stated to be unresponsive to glucagon, the investigators anticipate that the liver will be responsible, in part, for the increase in EGP.

ELIGIBILITY:
Inclusion Criteria:

* 25-35 kg/m^2
* Normal Glucose Tolerance subjects (24)
* Type 2 Diabetic Subjects (24)
* Diabetic subjects must be on a stable dose (more than 3 months) of monotherapy or combination therapy with metformin and/or a sulfonylurea
* Diabetic subjects must have HbA1c <8.0%
* Other than diabetes, subjects must be in good general health as determined by physical exam, medical history, blood chemistries, CBC (complete blood count), TSH (thyroid-stimulating hormone), T4 (thyroxine), EKG (electrocardiogram) and urinanalysis.
* Only subjects whose body weight has been stable (± 3 lbs) over the preceding three months and who do not participate in an excessively heavy exercise program will be included.

Exclusion Criteria:

* Subjects taking drugs known to affect glucose metabolism (other than metformin and sulfonylurea) will be excluded.
* Individuals with evidence of proliferative diabetic retinopathy, plasma creatinine >1.4 females or >1.5 males, or 24-hour urine albumin excretion > 300 mg will be excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-05-23 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2023-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eugenio Cersosimo, MD,PhD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- University of Texas Health Science Center, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | T2DM Individuals on Dapagliflozin | T2DM Individuals on Placebo | Normal Glucose Tolerance (NGT) on Dapagliflozin | Normal Glucose Tolerance (NGT) Placebo
Started | 13 | 7 | 8 | 4
Completed | 13 | 7 | 8 | 4
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | T2DM Individuals on Dapagliflozin | T2DM Individuals on Placebo | Normal Glucose Tolerance (NGT) on Dapagliflozin | Normal Glucose Tolerance (NGT) Placebo | Total
Number analyzed (Participants) | 13 | 7 | 8 | 4 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (3) | 58 (1.7) | 44 (2.2) | 47 (4.9) | 51.5 (2.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 13 | 7 | 8 | 4 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 6 | 1 | 14
  Not Hispanic or Latino | 9 | 4 | 2 | 3 | 18
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 0 | 2
  White | 12 | 7 | 7 | 4 | 30
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 7 | 8 | 4 | 32

OUTCOME MEASURES:

1. Primary Outcome: Endogenous Glucose Production Measurement
Description: Endogenous Glucose Production in NGT/T2DM subjects before and after dapagliflozin/Placebo administration from baseline to 240 minutes.
Time Frame: 3 weeks
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | T2DM Individuals on Dapagliflozin | T2DM Individuals on Placebo | Normal Glucose Tolerance (NGT) on Dapagliflozin | Normal Glucose Tolerance (NGT) Placebo
Number analyzed (Participants) | 13 | 7 | 8 | 4
mg/dl | 155 (6.4) | 121 (6.2) | 104 (4.2) | 98 (2)

2. Secondary Outcome: Renal Glucose Production Measurement of Change
Description: Renal Glucose Production in T2DM and NGT subjects before and after dapagliflozin/placebo administration from baseline to 240 minutes.
Time Frame: Baseline to 3 weeks
Measure: Mean (Standard Deviation); unit: mg/kg.min
Arm/Group | T2DM Individuals on Dapagliflozin | T2DM Individuals on Placebo | Normal Glucose Tolerance (NGT) on Dapagliflozin | Normal Glucose Tolerance (NGT) Placebo
Number analyzed (Participants) | 13 | 7 | 8 | 4
mg/kg.min
  Baseline | 0.09 (0.04) | 0.01 (0.03) | 0.03 (0.09) | 0.03 (0.09)
  3 weeks | 0.17 (0.05) | 0.03 (0.05) | 0.09 (0.1) | 0.14 (0.12)

ADVERSE EVENTS:
Time Frame: 4 years
Arm/Group | T2DM Individuals on Dapagliflozin | T2DM Individuals on Placebo | Normal Glucose Tolerance (NGT) on Dapagliflozin | Normal Glucose Tolerance (NGT) Placebo
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/7 | 0/8 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/7 | 0/8 | 0/4
Other Adverse Events (participants affected / at risk) | 0/13 | 1/7 | 1/8 | 0/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | T2DM Individuals on Dapagliflozin (N=13) | T2DM Individuals on Placebo (N=7) | Normal Glucose Tolerance (NGT) on Dapagliflozin (N=8) | Normal Glucose Tolerance (NGT) Placebo (N=4)
Transcient Syncope (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) — Participants had been lying in bed and got up too soon from the bed and felt dizzy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-18): https://cdn.clinicaltrials.gov/large-docs/66/NCT02981966/Prot_SAP_000.pdf